CLINICAL TRIAL: NCT07182214
Title: An Observational Study on the Assessment of Lung Cancer Using Liquid Biopsy for Collecting miRNA Expression Profile and DNA Methylation Biomarkers
Status: Recruiting | Type: Observational
Sponsor: Pharus Taiwan, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PHA-CPIP-LUN-A001
Record Dates: First submitted 2025-09-11; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- control/test: Participants in the test group must have identified lung nodules or masses through low-dose computed tomography (LDCT)CT scan, and have a scheduled medical operation, which is not limited to surgical excision. Control group participants should have no significant findings in LDCT/CT scan displaying either no nodules, or nodules smaller than 6mm were assessed by investigators without clinically significant justification.
  Interventions: Other: Collect blood sample

INTERVENTIONS:
Other: Collect blood sample — Collect venous blood sample from subjects prior fasting, any operation or treatment

SUMMARY:
The purpose of this study is to observe whether miRNA and DNA methylation collected through liquid biopsy can serve as a biomarker for evaluating lung cancer.

DETAILED DESCRIPTION:
The purpose of this study is to observe whether miRNA and DNA methylation collected through liquid biopsy can serve as a biomarker for evaluating lung cancer. Lung cancer is a highly prevalent and lethal cancer, ranking second among common cancers worldwide with approximately 2.21 million new cases reported in 2020, according to the World Health Organization (WHO). It also caused around 1.8 million deaths, making it the leading cause of cancer-related mortality. This trend is consistent at the national level as well. The American Cancer Society (ACS) estimates approximately 140,000 new cases of lung cancer in the United States in 2023, ranking second in incidence among common cancers and first in mortality, accounting for about one-fifth of all cancer deaths. In Taiwan, the latest statistical report from the Health Promotion Administration, Ministry of Health and Welfare (HPA) in 2020 shows that cases of lung, bronchus, and tracheal malignant tumors accounted for 13.42% of all malignant tumor cases, totaling 16,360 individuals, ranking second in incidence for both males and females and first in mortality.

Similar to most cancers, early detection of lung cancer and timely treatment can improve survival rates. Low-dose computed tomography (LDCT) is currently an internationally recognized tool for early lung cancer screening, but it has a high false-positive rate of up to 95%, leading to overdiagnosis and causing anxiety in patients waiting for diagnosis results. Furthermore, confirmatory diagnosis of lung cancer often requires surgery or biopsy, with a rate of benign cases ranging from 10% to 30% among surgical patients. Overdiagnosis leads to the waste of healthcare resources and exposes healthy individuals to unnecessary surgical risks. Therefore, if there are other effective interventions available, it would provide physicians with additional tools to evaluate lung cancer and make decisions. These interventions could include positron emission tomography (PET) or potential methods that have not yet become routine tests, such as miRNA, DNA methylation, or circulating tumor DNA (ctDNA). This study will focus on miRNA to determine if it can assist in the evaluation of lung cancer.

This clinical study is a non-randomized, non-blinded, two-arm design trial. The participants (study subjects) in test group will be individuals at least 18 years old, and have been screened for lung nodules or masses using low dose computed tomography (LDCT)/CT scan and are scheduled for an operation (not limiting to surgical excision). Subjects in the control group will be individuals who are also at least 18 years old and have had a recent LDCT/CT scan with an axial resolution of 3 mm or less, showing no significant findings displaying either no nodules, or nodules smaller than 6mm were assessed by investigators without clinically significant justification, within 2 months prior to the enrollment for this study. Real-time polymerase chain reaction (RT-qPCR) and next-generation sequencing (NGS) techniques will be employed to detect the expression profile of miRNA and DNA methylation in plasma. Tumor marker test results and relevant information will be collected for analysis, with post operation biopsy results or physician judgments based on medical images tracked within 2 months serving as the standard for evaluating the effectiveness of lung cancer assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male participants at least 18 years of age
2. Participants in the test group must have identified lung nodules or masses through low-dose computed tomography (LDCT)CT scan, and have a scheduled medical operation, which is not limited to surgical excision. Control group participants should have no significant findings in LDCT/CT scan displaying either no nodules, or nodules smaller than 6mm were assessed by investigators without clinically significant justification, through an axial resolution of 3 mm or less, within 2 months prior to their enrollment in the study.
3. Participants in the test group should be treatment naïve.
4. Ability to complete a questionnaire, comprehend and comply with the requirements of the study
5. Written informed consent, and authorization to use and disclose health information

Exclusion Criteria:

1. Has any history of cancer diagnosis
2. Has received a blood transfusion (except for autologous blood transfusion) within the first two months prior to participating the trial
3. Is participating in a clinical trial (the non-intervention trial will be accepted)
4. Has taken gene therapy within one year prior to participating the trial
5. Has any vaccinations within 3 months prior to blood sample collection
6. Is currently pregnant
7. Has any severe acute or uncontrolled chronic lung disease such as pneumonia, lung abscess, acute exacerbation of COPD or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of Study results and, in the judgment of the Investigator, would make the patient inappropriate for entry into this Study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants in the test group must have identified lung nodules or masses through low-dose computed tomography (LDCT)CT scan, and have a scheduled medical operation, which is not limited to surgical excision. Control group participants should have no significant findings in LDCT/CT scan displaying either no nodules, or nodules smaller than 6mm were assessed by investigators without clinically significant justification, through an axial resolution of 3 mm or less, within 2 months prior to their enrollment in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1340 (Estimated)
Dates: Start 2024-05-05 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To observe miRNA or DNA methylation expressions between subjects with and without lung cancers. Once the primary outcome has been reached and the hypothesis has proven true for this study, study team then will evaluate for the secondary outcome. | 1-56 days

CONTACTS AND LOCATIONS:
Locations (1):
- Pharus Taiwan, Inc., Hsinchu, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided